CLINICAL TRIAL: NCT07347795
Title: Blood Flow Restriction Training and Hand Grip Strength in Hemiparetic CP
Brief Title: Effect of Blood Flow Restriction Training Exercises on Hand Grip Strength in Hemiparetic Cerebral Palsied Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Saeed Alsakhawi, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005952
Record Dates: First submitted 2025-12-31; First posted 2026-01-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy Spastic Hemiplegic
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group performs traditional hand grip strengthening exercises, focusing on similar exercises but without blood flow restriction. Both groups participate in a similar frequency and duration of training, with a gradual increase in repetitions over the 8 weeks
  Interventions: Behavioral: control group
- Study group (Experimental)
  Interventions: Device: Blood Flow Restriction Training Exercises group

INTERVENTIONS:
Device: Blood Flow Restriction Training Exercises group — The BFR group underwent BFR training for 8 weeks, with sessions held three times per week. A tourniquet-style cuff is placed on the upper arm to restrict blood flow during exercise. The exercises involved are low-intensity grip strengthening activities (e.g., squeezing a rubber ball, gripping a hand dynamometer) at 20% of their one-repetition maximum (1RM). The cuff pressure is set at 50-70% of the participants' limb occlusion pressure, as determined by an initial assessment.
  Arms: Study group
Behavioral: control group — The control group performs traditional hand grip strengthening exercises, focusing on similar exercises but without blood flow restriction. Both groups participate in a similar frequency and duration of training, with a gradual increase in repetitions over the 8 weeks.
  Arms: Control group

SUMMARY:
The study aims to investigate the effect of blood flow restriction (BFR) training exercises on the hand grip strength of children with hemiparetic cerebral palsy. Hand grip strength is a vital component of motor function and is often severely compromised in children with hemiparetic CP, which can significantly impact their daily activities and quality of life. Blood flow restriction (BFR) training is a novel exercise technique where a cuff or band is used to partially occlude blood flow during low-intensity resistance exercises. This method has been shown to stimulate muscle growth and strength gains similar to those achieved through high-intensity strength training, without the need for high loads. Given the unique physiological challenges faced by children with hemiparetic CP, BFR training could provide an effective alternative to traditional strength training methods.

ELIGIBILITY:
Inclusion Criteria:

Age will range from 6-12 years

* Diagnosed with hemiparetic cerebral palsy (right or left side).
* According to Modified Ashwer scale, has grade 1 or 1+ grade
* Children with the ability to understand and follow verbal commands and instructions used during training and tests

Exclusion Criteria:

* Any contraindications to exercise, such as moderate or severe spasticity, orthopedic deformities, or other serious health conditions.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength measured using a handheld dynamometer | 8 weeks
  Hand grip strength of the affected hand will be assessed using a calibrated handheld dynamometer. The maximum voluntary grip force will be recorded in kilograms (kg). Three trials will be performed, and the highest value will be used for analysis.
muscle thickness at the midpoint of the forearm flexor muscles | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Universit, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No